CLINICAL TRIAL: NCT06570109
Title: Association Between Decline in Functional Ability and Frailty in Community-dwelling Older Adults Living With Alzheimer's Dementia
Brief Title: Frailty Outcomes And Risk With Alzheimer's Related Dementia
Acronym: FORWARD
Status: Enrolling by invitation | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Riis, MD, Aalborg University Hospital
Other Study IDs: N-20230068
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail: Defined by Fried Frailty Criteria
  Interventions: Other: Frailty
- Non-Frail/pre-frail: Defined by Fried Frailty Criteria

INTERVENTIONS:
Other: Frailty — defined as weigh loss (>4.5 kg in one year), exhaustion, slow gait speed (below 20th percentile for sex and height), weakness (handgrip strength below 20th percentile for sex and BMI), and low physical activity (by the Physical Activity Scale for the Elderly). The presence of three or more out of five criteria is defined as frailty while one to two criteria is prefrailty
  Groups: Frail

SUMMARY:
The primary aim of this study is to investigate the association between frailty as defined by the Fried Frailty Phenotype and risk of functional decline in patients with Alzheimer's dementia. The hypothesis is that frailty is associated with greater functional decline in community-dwelling older people with Alzheimer's dementia compared to those without frailty.

Secondary aims include investigation of long-term risk of institutionalization (through administrative follow-up) and trajectories of assessment components in future assessment.

The study is designed as a prospective cohort study. Participants in the study will undergo an assessment battery at baseline, 1 years of follow-up, and administrative follow-up for 5 years.

Participants will be recruited from patients of the Unit of Dementia at Aalborg University Hospital within 3 months of dementia diagnosis. The time frame of 3 months after diagnosis was chosen to ensure that cognitive assessment in the Unit of Dementia was reflective of patient's cognitive level and thereby ability to consent at inclusion. Patients will be eligible for inclusion if they are 65 years or older, have a diagnosis of mild or moderate Alzheimer's or mixed (Alzheimer's and vascular) dementia, live at home, and are able to walk 5 meters independently of other people (walking aids will be allowed). The severity of dementia will be defined according to score on the Mini Mental State Examination (MMSE) as it has done in other studies. According to this definition a MMSE score between 20-30 indicates mild Alzheimer's dementia and a MMSE score from 15-19 indicates moderate dementia. People with moderately severe and severe Alzheimer's dementia defined as MMSE score below 15 will not be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimers Dementia
* MMSE > 14
* Age >= 65
* Not living in institution
* Able to walk 5m without assistence (walking aids accepted)

Exclusion Criteria:

* No available caregiver/proxy
* Unable to give informed consent as judged by caregiver/proxy or researcher
* Time from diagnosis > 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study aims to include community-dwelling people living at home with mild to moderate Alzheimers dementia aged 65+. Participant will be included only within 3 months of dementia diagnosis. Consecutive sampling at the Unit of Dementia in Northen Jutland in Denmark will be employed.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Caregiver IADL Change | 1 year
  Defined by caregiver reported ADL performance on the Functional Activities Questinnaire
Patient IADL Change | 1 year
  Defined by patient reported ADL performance on the Functional Activities Questinnaire
Caregiver BADL Change | 1 year
  Defined by caregiver reported ADL performance on Barthel ADL scale
Patient BADL Change | 1 year
  Defined by patient reported ADL performance on Barthel ADL scale

SECONDARY OUTCOMES:
Nursing home admission | 5 years
  Admission to nursing home (time to event)
Mortality | 5 years
  Death (time to event)

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT06570109/SAP_000.pdf